CLINICAL TRIAL: NCT01675739
Title: Effectiveness of Fixed Preparation-to-Colonoscopy Interval Using Short Message Service (SMS) for Afternoon Colonoscopy: a Randomized Control Study
Brief Title: Effectiveness of Fixed PC Interval Using SMS for Afternoon Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jongha Park, Assistant professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SMS-CFS
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Effectiveness of SMS to Fix PC Interval
Keywords: colonoscopy; bowel preparation; short message service
MeSH Terms: interventions — Polyethylene Glycols; Golytely

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- No-SMS group (Active Comparator): In No-SMS group took 1st 2L of PEG solution at 6-8 PM on the day before colonoscopy and started drinking the 2nd 2L PEG at about 6hours before the day of the colonoscopy without SMS.
  Interventions: Drug: polyethylene glycol (PEG)
- SMS group (Experimental): Patients in SMS group took 1st 2L PEG as same manner of No-SMS group and then started drinking the 2nd 2L PEG at about 6hours before the day of the colonoscopy after receiving scheduled short message service(SMS)
  Interventions: Behavioral: Short message service of mobile phone (SMS); Drug: polyethylene glycol (PEG)

INTERVENTIONS:
Behavioral: Short message service of mobile phone (SMS) — In SMS group, patients took 1st dose polyethylene glycol (PEG) 2L at 6-8pm the day before colonoscopy and then start to take 2nd dose PEG 2L after receiving Short message service of mobile phone (SMS) 6hours before afternoon colonoscopy.
  Arms: SMS group
Drug: polyethylene glycol (PEG) — No-SMS group took 1st 2L of PEG solution at 6-8 PM on the day before colonoscopy and started drinking the 2nd 2L PEG at about 6hours before the day of the colonoscopy.
  SMS group took 1st 2L PEG as same manner of No-SMS group and then started drinking the 2nd 2L PEG at about 6hours before the day of the colonoscopy after receiving scheduled SMS
  Other Names: Colyte

SUMMARY:
The purpose of this study is to evaluate the effectiveness of SMS (short message service of mobile phone) reminder to fix PC interval for bowel preparation in afternoon colonoscopy.

DETAILED DESCRIPTION:
Bowel preparation quality for colonoscopy is influenced by several factors and preparation-to-colonoscopy (PC) interval is one of the important factors. The bowel preparation with split-dose PEG (polyethylene glycol) is an obviously uncomfortable process, it is usually difficult to ingest PEG in time. Therefore, the investigators conducted a prospective randomized control study to evaluate the effectiveness of fixed PC interval for satisfactory bowel preparation in the afternoon colonoscopy using mobile phone short message service (SMS), which reported that it could increase patient's compliance in other practical era

ELIGIBILITY:
Inclusion Criteria:

* 18 and 80 years who were scheduled for afternoon colonoscopy (screening or surveillance)

Exclusion Criteria:

* unavailable mobile phone nor SMS
* age younger than 18 years
* pregnancy
* breastfeeding
* history of large-bowel resection
* renal failure (serum creatinine ≥ 3.0 mg/dL [normal 0.8-1.4])
* drug addiction or major psychiatric illness
* allergy to PEG
* refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
the Ottawa bowel preparation scale | at the end of time of the colonoscopic examination (about 30 minutes-1hour)
  This scale assesses cleanliness and fluid volume respectively and presents the total score as sum of these two values. Cleanliness was assessed for the right colon (cecum, ascending colon), midcolon (transverse, descending colon), and the rectosigmoid colon; each colon section was individually rated from 0 to 4 (0 = no liquid, 1 = minimal liquid, no suction required, 2 = suction required to see mucosa, 3 = wash and suction required, 4 = solid stool, not washable). Fluid quantity was rated from 0 to 2 for the entire colon (0 = minimal, 1 = moderate, 2 = large). The Ottawa Scale scores range from 0 (perfect) to 14 (solid stool in each colon segment and large amount of fluid).

CONTACTS AND LOCATIONS:
Overall Officials: Tae Oh Kim, Principal Investigator — Department of Internal Medicine, Haeundae Paik Hospital, Inje University, College of Medicine
Locations (1):
- Department of Internal Medicine, Haeundae Paik Hospital, Inje University, College of Medicine, Busan, South Korea